CLINICAL TRIAL: NCT06038578
Title: A Randomized, Multicenter, Open-Label, Phase 2 Study of TRK-950 When Used in Combination With Ramucirumab and Paclitaxel in Patients With Gastric Cancer
Brief Title: A Study of TRK-950 When Used in Combination With Ramucirumab and Paclitaxel in Patients With Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 950GCV01
Record Dates: First submitted 2023-08-29; First posted 2023-09-15 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: Gastric Cancer, Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; TRK-950; CAPRIN-1
MeSH Terms: conditions — Stomach Neoplasms; Adenocarcinoma | interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm A: TRK-950(5 mg/kg)+Ramucirumab+Paclitaxel (Experimental): Participants who will be randomized to receive a 5 mg/kg intravenous(IV) dose of TRK-950 on days 1, 8, 15 and 22 in combination with 8 mg/kg IV dose of ramucirumab on days 1 and 15 and 80 mg/m^2 IV dose of paclitaxel on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Biological: TRK-950; Drug: Ramucirumab; Drug: Paclitaxel
- Arm B: TRK-950(10 mg/kg)+Ramucirumab+Paclitaxel (Experimental): Participants who will be randomized to receive a 10 mg/kg intravenous(IV) dose of TRK-950 on days 1, 8, 15 and 22 in combination with 8 mg/kg IV dose of ramucirumab on days 1 and 15 and 80 mg/m^2 IV dose of paclitaxel on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Biological: TRK-950; Drug: Ramucirumab; Drug: Paclitaxel
- Arm C: Ramucirumab+Paclitaxel (Active Comparator): Participants who will be randomized to receive a 8 mg/kg IV dose of ramucirumab on Days 1 and 15 in combination with 80 mg/m^2 IV dose of paclitaxel on Days 1, 8, and 15 of a 28-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Biological: TRK-950 — 5 mg/kg or 10 mg/kg IV infusion over 60 minutes on Day 1, 8, 15 and 21 of each 28 day cycle
  Arms: Arm A: TRK-950(5 mg/kg)+Ramucirumab+Paclitaxel; Arm B: TRK-950(10 mg/kg)+Ramucirumab+Paclitaxel
Drug: Ramucirumab — 8 mg/kg IV infusion on Days 1 and 15 of a 28-day cycle
  Other Names: CYRAMZA®
Drug: Paclitaxel — 80 mg/m^2 IV infusion on Days 1, 8, and 15 of a 28-day cycle

SUMMARY:
This study will assess the efficacy, safety, optimal dose and ADA and NAbs development of TRK-950 at two separate dose levels in combination with ramucirumab and paclitaxel (RAM+PTX) as compared with RAM + PTX treatment alone in participants with gastric or gastro-esophageal junction (GEJ) adenocarcinoma.

DETAILED DESCRIPTION:
This study will assess and compare the efficacy, safety, pharmacokinetics (PK), optimal dose and anti-drug antibodies (ADA) and neutralizing antibodies (NAbs) development of TRK-950 at two separate dose levels in combination with RAM + PTX as compared with RAM + PTX treatment alone in participants with gastric or gastro-esophageal junction (GEJ) adenocarcinoma. The primary objective is progression free survival (PFS). Secondary objectives are overall survival, objective response rate, best overall response, duration of response, disease control rate, safety, pharmacokinetics, and immunogenicity of TRK-950 when used in combination with RAM+PTX.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic, or locally advanced and unresectable gastric or GEJ adenocarcinoma.
* The patient is eligible to receive Ramucirumab + Paclitaxel.
* Documented objective radiographic or clinical disease progression (e.g., any new or worsening malignant effusion documented by ultrasound examination) which may be confirmed by pathologic criteria (histology and/or cytology) if appropriate, during or after treatment. The prior treatment must meet one of the following criteria with the following treatment history:

  1. First treatment for metastatic disease or locally advanced disease without experiencing adjuvant / neo-adjuvant treatment, which progressed during treatment or within 4 months after the last dose of treatment
  2. Adjuvant / neo-adjuvant treatment which progressed more than 6 months after the last dose of treatment and first treatment for metastatic disease or locally advanced disease, which progressed during the treatment or within 4 months after the last dose of treatment
  3. Adjuvant / neo-adjuvant treatment which progressed during treatment or within 6 months after the last dose of treatment
  4. Adjuvant / neo-adjuvant treatment which progressed during treatment or within 6 months after the last dose of treatment and first treatment for metastatic disease or locally advanced disease, which progressed during treatment or within 4 months after the last dose of treatment
* Presence of primary or metastatic disease, measurable per RECIST v1.1 on CT scan.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Life expectancy of at least 3 months.
* Age ≥ 18 years in the US and Japan, and ≥ 19 years of age in Korea.
* Signed, written IRB-approved informed consent.
* Adequate organ function from specimens collected within 14 days prior to Day 1.
* For men and women of child-producing potential, the use of effective contraceptive methods during the study and for 6 months after the last dose of TRK-950.
* All patients must sign a pre-screening consent to assess tumor tissue to determine eligibility. Tumor tissue must be evaluable for CAPRIN-1 staining at a CLIA certified laboratory and meet or exceed the cutoff value (30% at ≥ 2+ staining) as defined in the expression level requirements.

Exclusion Criteria:

* Prior history of treatment with ramucirumab or paclitaxel.
* HER2 positive gastric or GEJ adenocarcinoma.
* Major surgery within 28 days prior to randomization.
* Baseline corrected QT (QTc) interval of > 470 msec for females and > 450 msec for males calculated using Fridericia's formula.
* New York Heart Association (NYHA) Class II - IV symptomatic congestive heart failure, or symptomatic or poorly controlled cardiac arrhythmia.
* The patient has experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 3 months prior to randomization.
* The patient has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Clinically symptomatic venous thromboembolism or current treatment with anti-coagulants. (Patients receiving prophylactic and low-dose anticoagulation therapy are eligible provided that the coagulation parameter defined in the Inclusion Criterion 9 is met.)
* Uncontrolled arterial hypertension ≥ 150 mmHg (systolic) or ≥ 90 mmHg (diastolic) despite standard medical management.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Pregnant or nursing women.
* Treatment with radiation therapy within 2 weeks, or treatment with chemotherapy, immunotherapy, targeted therapy, or investigational therapy within 4 weeks prior to randomization (within 2 weeks for Oral FU (S1 and capecitabine)).
* The patient has significant bleeding disorders, vasculitis, or had a significant bleeding episode from the gastrointestinal tract within 3 months prior to randomization.
* Clinically significant ascites, paracentesis in the last 3 months, or undergoes regular paracentesis procedures.
* History of gastrointestinal perforation and/or fistulae within 6 months prior to randomization.
* The patient has a serious or non-healing wound, peptic ulcer, or bone fracture within 28 days prior to randomization.
* The patient has a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (e.g., hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Known active infection with HIV, hepatitis B or hepatitis C. Patients with a history of hepatitis B or C are allowed if HBV DNA or Hep C RNA are undetectable.
* The patient is currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study. Patients who have recently discontinued dosing of study drug are eligible to participate as long as the final dose of study drug was ≥ 28 days from randomization for participation in this study. Patients participating in surveys or observational studies are eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival (PFS) | Time from date of randomization to the date of progressive disease or death due to any cause, whichever occurs first, up to approximately 24 months
  Progression free Survival (PFS) is defined as time from the date of randomization to the date of progressive disease or death due to any cause based on Independent Central Review.

SECONDARY OUTCOMES:
Overall survival (OS) | Time from the date of randomization to the date of death due to any cause, up to approximately 24 months
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
Objective response rate (ORR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  Objective response rate (ORR) is defined as the proportion of participants who achieve a best overall response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Independent Central Review.
Progression free Survival (PFS) | Time from date of randomization to the date of progressive disease or death due to any cause, whichever occurs first, up to approximately 24 months
  Progression free Survival (PFS) is defined as time from the date of randomization to the date of progressive disease or death due to any cause based on investigator assessment.
Objective response rate (ORR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  Objective response rate (ORR) is defined as the proportion of participants who achieve a best overall response of complete response (CR) or partial response (PR) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by investigator.
Best overall response (BOR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  The best overall response is defined as the best overall response (BOR) recorded from the start of treatment until the end of treatment and includes CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Independent Central Review based.
Best overall response (BOR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  The best overall response is defined as the best overall response (BOR) recorded from the start of treatment until the end of treatment and includes CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE) using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by investigator.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  Disease control rate (DCR) is defined as the proportion of participants who achieve a best overall response of complete response (CR), partial response (PR) or stable disease (SD) for a minimum of 6 weeks using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by Independent Central Review based.
Disease control rate (DCR) | From start of treatment to date of documented disease progression, up to approximately 24 months
  Disease control rate (DCR) is defined as the proportion of participants who achieve a best overall response of complete response (CR), partial response (PR) or stable disease (SD) for a minimum of 6 weeks using the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria as assessed by investigator.
Duration of response (DoR) | Time from initial response (CR or PR) to date of documented disease progression or death due to any cause, whichever occurs first, up to approximately 24 months
  Duration of response (DoR) is defined as the time from the initial response (CR or PR) until documented tumor progression or death from any cause based on Independent Central Review based.
Duration of response (DoR) | Time from initial response (CR or PR) to date of documented disease progression or death due to any cause, whichever occurs first, up to approximately 24 months
  Duration of response (DoR) is defined as the time from the initial response (CR or PR) until documented tumor progression or death from any cause based on investigator assessment.
Incidence of Treatment-emergent Adverse Events (TEAE) | From time subjects are enrolled up to 45 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Serious Adverse Events (SAEs) | From time subjects are enrolled up to 45 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Adverse Events of Special Interest (AESI) | From time subjects are enrolled up to 45 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Incidence of Discontinuation due to AE | From time subjects are enrolled up to 45 days after last study dose
  Adverse events will be graded according to the National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0.
Incidence of Physical Examination Findings, Vital sign measurements, Standard clinical laboratory parameters, ECG parameters | From time subjects signs informed consent form up to 45 days after last study dose
Pharmacokinetic Parameter of Concentration of drug at the end of infusion (CEOI) of TRK-950 | Cycle 1 on day 1 and 15, subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Trough Serum Concentration (Ctrough) of TRK-950 | Cycle 1 on day 1 and 15, subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Area Under the Curve (AUC) of TRK-950 | Cycle 1 on day 1 and 15, subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Concentration of drug at the end of infusion (CEOI) of Ramucirumab | Cycle 1 and 4 on day 1 and 15, Cycles 2, 3 and subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Trough Serum Concentration (Ctrough) of Ramucirumab | Cycle 1 and 4 on day 1 and 15, Cycles 2, 3 and subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Area Under the Curve (AUC) of Ramucirumab | Cycle 1 and 4 on day 1 and 15, Cycles 2, 3 and subsequent cycles on day 1 (each cycle is 28 days)
Pharmacokinetic Parameter of Concentration of drug at the end of infusion (CEOI) of Paclitaxel | Cycle 1 and 4 on day 1 and 15 (each cycle is 28 days)
Pharmacokinetic Parameter of Trough Serum Concentration (Ctrough) of Paclitaxel | Cycle 1 and 4 on day 1 and 15 (each cycle is 28 days)
Pharmacokinetic Parameter of Area Under the Curve (AUC) of Paclitaxel | Cycle 1 and 4 on day 1 and 15 (each cycle is 28 days)
Percentage of participants who are Anti-drug antibody (ADA)-Positive and Neutralizing antibodies (NAbs) | Cycle 1 on day 1 and 15, subsequent cycles on day 1 (each cycle is 28 days)
Change from Baseline in Patient Reported Quality of Life assessed by the Questionnaire - Core questionnaire EORTC QLQ-C30 scores | From Cycle 1 on day 1 through study completion, up to approximately 24 months (each cycle is 28days)
  The EORTC QLQ-C30 consists of 30 questions assessing global health-related quality of life for cancer patients. It incorporates five functional scale (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), and six single-items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change from Baseline in Patient Reported Quality of Life assessed by Questionnaire - EuroQOL Five Dimensions questionnaire 3L (EQ-5D-3L) scores | From Cycle 1 on day 1 through study completion, up to approximately 24 months (each cycle is 28days)
  The EQ-5D questionnaire consists of the following five dimensions, each describing a different aspect of health: Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety/ Depression. The participants self-assess each dimension has three response levels of severity: no problems, some problems, extreme problems.

CONTACTS AND LOCATIONS:
Locations (27):
- United States (14):
  - City of Hope, Duarte, California
  - City of Hope at Orange County Lennar Foundation Cancer Center, Irvine, California
  - University of California, Los Angeles, Santa Monica, California
  - Texas Oncology Arlington North, Arlington, Texas
  - Texas Oncology Bedford, Bedford, Texas
  - Texas Oncology Dallas Methodist, Dallas, Texas
  - Texas Oncology Dallas Medical City, Dallas, Texas
  - Texas Oncology Dallas Presbyterian, Dallas, Texas
  - Texas Oncology Methodist Charlton Cancer Center, Dallas, Texas
  - Texas Oncology-Sammons Cancer Center, Dallas, Texas
  - Texas Oncology Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology Grapevine, Grapevine, Texas
  - Texas Oncology Plano East, Plano, Texas
  - Texas Oncology Plano West, Plano, Texas
- Japan (7):
  - Kanagawa Prefectural Hospital Organization Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saitama Prefectural Hospital Organization Saitama Cancer Center, Shinden, Saitama
  - Shizuoka Cancer Center, Nagaizumi-cho, Shizuoka
  - National Cancer Center Hospital, Chūōku
  - Osaka International Cancer Institute, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtoku
- South Korea (6):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Severance Hospital, Seoul
  - ASAN Medical Center, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No